CLINICAL TRIAL: NCT04149834
Title: Clinical and Radiographic Evaluation of Non-Incised Papilla Surgical Approach Versus Modified Minimally Invasive Surgical Technique in Treatment of Intra-osseous Defects in Patients With Stage III Periodontitis: A Randomized Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of NIPSA Versus M-MIST in Treatment of Intra-osseous Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa EL-Desouky Helal, Lecturer assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PER3-3-2
Record Dates: First submitted 2019-10-20; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Periodontitis, Adult
Keywords: Intraossous defects; Periodontitis
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis

STUDY DESIGN:
Intervention Model Description: • The patients will be randomly assigned into two groups: Group A (Test): Patients will receive Non-Incised Papilla Surgical Approach (NIPSA)
  • Group B (Control): Patients will receive Modified Minimally Invasive Surgical technique (M-MIST)
Masking Description: Single blinded:
  * Blinding of the participants is not applicable.
  * Blinding of the operator is not applicable.
  * Outcome assessor (primary and secondary outcomes) & biostatistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Minimally Invasive Surgical Technique (Active Comparator): Comparator: Modified Minimally Invasive Surgical Technique The defect will be gained through the tiny buccal triangular ﬂap: from the buccal 'window' the soft tissue ﬁlling the defect (i.e. the so-called granulation tissue) will be sharply dissected from the papillary supra-crestal connective tissue and from the bony walls with a micro-blade and will be removed with a mini-curette (The soft tissue will be sharply dissected from the osseous defect)
  Interventions: Procedure: Group B (Control): Patients will receive M-MIST
- Non- incised papilla surgical approach (Other): intervention: Non- incised papilla surgical approach Apical horizontal incision on the buccal mucosa, as far as possible from the interdental papillae and marginal KT will be performed. Soft tissue will be reflected apico-coronally by a full-thickness flap showing the granulation tissue filling the bony defect after exposing the coronal limit of the intra-bony component of the defect, while the marginal tissue will be kept unaltered.
  Interventions: Procedure: Group A (Test): Patients will receive NIPSA

INTERVENTIONS:
Procedure: Group A (Test): Patients will receive NIPSA — patients received Non- incised papilla surgical approache
  Arms: Non- incised papilla surgical approach
Procedure: Group B (Control): Patients will receive M-MIST — patients received Modified Minimally Invasive Surgical Technique
  Arms: Modified Minimally Invasive Surgical Technique

SUMMARY:
The aim: Clinical and Radiographic Evaluation for intra-osseous defects in stage III periodontitis using NIPSA versus M-MIST Steps in short Pre-surgical therapy

• Before surgical intervention, each patient will be given careful instructions on proper oral hygiene measures.

Surgical Procedures:

* Group B (Control): Patients will receive Modified Minimally Invasive Surgical technique (M-MIST) Group A (Test): Patients will receive Non-Incised Papilla Surgical Approach (NIPSA) Postoperative medication
* Administration of amoxicillin (500 mg tabs) T.I.D for 7 days and Metronidazole (500 mg tabs) T.I.D for 7 days
* Rinsing with Chlorhexidine 0.12% (B.I.D for 14 days).
* Ibuprofen 600 mg tabs once every 8h could be administrated in case of unbearable pain
* Follow up period: after 8 weeks/ after surgery by 1 week- 1 month- 3 months- 6 months- 1 year

DETAILED DESCRIPTION:
P: Population: Stage III periodontitis presenting intraosseous defects I: Intervention: Non-Incised Papilla Surgical Approach (NIPSA) C: Control: Modified Minimally Invasive Surgical Technique (M-MIST) O: Outcome measurements T: 1- year S: Randomized clinical trial

Surgical Procedures:

The operator will anesthetize the surgical sites with 4% ARTINIBSA containing Articaine hydrochloride Epinephrine (adrenaline) 1: 100.000 injection for both groups. For patients that recieved (NIPSA) as reported by (Moreno Rodríguez and Caffesse 2017).

* After locally anesthetizing the area an apical horizontal incision on the buccal mucosa, as far as possible from the interdental papillae and marginal KT will be performed. Soft tissue will be reflected apico-coronally by a full-thickness flap showing the granulation tissue filling the bony defect after exposing the coronal limit of the intra-bony component of the defect, while the marginal tissue will be kept unaltered.
* Horizontal mattress sutures with single interrupted sutures will be placed as the second line of closure.

while patients that received (M-MIST) reported by (Banthia et al. 2016a)

* Access to the defect will be gained through the tiny buccal triangular ﬂap: from the buccal 'window' the soft tissue ﬁlling the defect (i.e. the so-called granulation tissue) will be sharply dissected from the papillary supra-crestal connective tissue and from the bony walls with a micro-blade and will be removed with a mini-curette (The soft tissue will be sharply dissected from the osseous defect)
* No interdental and/or lingual intra-sulcular incisions will be performed. The supra-crestal interdental tissues.
* Surgical flaps will be sutured to the pre-surgical level with 5-0 vicryl suture utilizing single interrupted suturing techniques that will achieve primary closure.
* Sutures will be removed 2 weeks post-surgically. Patients will be asked to discontinue mechanical tooth-brushing technique in the surgical area for 2 weeks.
* After this period, patients will be instructed to continue mechanical tooth brushing again of the treated sites using a soft toothbrush.

Patients will be recalled monthly for supportive periodontal therapy during the course of the study. And then will be recalled every six months for supportive periodontal therapy after the study.

ELIGIBILITY:
Inclusion Criteria:

* Stage III periodontitis patient having at least one tooth with Two walls or combined 2- to 3-walls intraosseous defects ≥ 3 mm deep (assessed by trans-gingival probing, radiographic examination) with clinical attachment level (CAL) ≥ 5mm and pocket depth (PD) ≥ 6 mm.
* Defect not extended to a root furcation area.
* Vital teeth
* Non-smokers.
* No history of intake of antibiotics or other medications affecting the periodontium in the previous 6 months.
* No periodontal therapy carried out in the past 6 months.
* Able to sign an informed consent form.
* Patients age between 20 and 60 years old.
* Patients who are cooperative, motivated, and hygiene conscious.
* Able to come for the follow up appointment's needed.
* Systemically free according to Modified Cornell Medical Index health questionnaire (Kark et al., 1964).

Exclusion Criteria:

* Pregnancy or breast feeding.
* The presence of an orthodontic appliance.
* Teeth mobility greater than grade I.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of CAL gain | baseline/ after 6 months & 1 year post-surgical
  Clinical attachment Level gain (CAL) by UNC Periodontal probe (mm)

SECONDARY OUTCOMES:
Assessment of PD reduction | 1 year
  UNC Perioodntal probe (mm)
gingival recession | 1 year
  UNC Perioodntal probe (mm)
radiographic bone fill. | 1 year
  Linear measurements standardized periapical radiograph (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo Unv, Cairo, Egypt